CLINICAL TRIAL: NCT05696899
Title: Determining the Efficacy of Essential Oil Aromatherapy in Children Undergoing Port Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Annette Nasr, Nurse Scientist Nursing Research and Evidence-Based Practice, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-68138; PEDSVAR0068 (Other: OnCore)
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Anxiety and Fear; Pain
Keywords: Aromatherapy; Port-a-Cath; Pediatric
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy (Experimental): Patients will be given STILL QuickTAB Medipack blended scent aromatherapy in addition to standard supportive measures, which include numbing cream, Child Life support, distraction, caregiver hold, or any combination of these, based on patient preference.
  Interventions: Other: STILL QuickTAB Medipack blended scent aromatherapy, manufactured by Soothing Scents
- Control Group (No Intervention): Participants will be offered standard supportive measures, which include numbing cream, Child Life support, distraction, caregiver hold, or any combination of these, based on patient preference.

INTERVENTIONS:
Other: STILL QuickTAB Medipack blended scent aromatherapy, manufactured by Soothing Scents — A resealable quick-tab dispenser with the 'therapeutic inhaled essential oils' lavender, bergamot, sweet orange, and ylang ylang.
  Arms: Aromatherapy

SUMMARY:
The purpose of this study is to determine if the use of aromatherapy impacts patient anxiety and pain scores surrounding port access in pediatric oncology patients between the ages of 4 years and 18 years.

DETAILED DESCRIPTION:
Specific aims include the following:

Aim 1: To compare pre and post port access anxiety scores for both control and intervention groups.

Aim 2: To assess pre and post port pain scores surrounding port access for both control and intervention groups.

Aim 3: To compare pain and anxiety scores between age groups. The overall goal of this pilot study is to identify if aromatherapy, using non-topical, STILL QuickTAB Medipack blended scent aromatherapy, manufactured by Soothing Scents, is effective as a valid non-pharmacologic supplementation in reducing anxiety and pain scores during port access in pediatric oncology patients.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 4 years and 18 years
2. Scheduled for port access with or without lab draw
3. Oncology, neuro-oncology, and stem cell transplant patients

Exclusion Criteria:

1. has asthma, reactive airway disease, or allergies to any of the ingredients we are using in the aromatherapy study (lavender, bergamot, sweet orange, and ylang ylang)
2. currently uses aromatherapy for port accesses or other painful procedures (does not apply to patients using aromatherapy, such as peppermint oil, for nausea)
3. has a cognitive impairment that prevents them from being able to provide anxiety or pain scores
4. does not wish to participate in the study

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Effect of aromatherapy on post patient anxiety scores | 5 minutes
  Comparison of pre and post patient anxiety scores for both control and intervention groups using the Visual Facial Anxiety Scale with corresponding values ranging from 0-10. 0 indicates no anxiety and 10 indicates the highest level of anxiety.
  Anxiety score will be measured by using the Visual Facial Anxiety Scale (VFAS)

SECONDARY OUTCOMES:
Effect of aromatherapy on post patient port pain scores | up to 7 minutes
  Comparison of pre and post patient pain scale for both control and intervention groups using the 0-10 scale or the Wong-Baker FACES Pain Rating Scale, according to patient preference and age appropriate rating. The Wong-Baker FACES Pain Rating Scale has corresponding faces for numerical rankings of 0-10. For both pain scales, 0 indicates no pain and 10 indicates the worst pain.

OTHER OUTCOMES:
Aromatherapy effect according to age | up to 7 minutes
  To compare pre and post pain and anxiety scores between the three age groups. The Visual Facial Anxiety Scale will be used to score patient anxiety, with faces corresponding to numerical ratings of 0-10. 0 corresponds with no anxiety and 10 corresponds with the highest level of anxiety. Pain will be scored using the 0-10 Numerical Rating Scale or the Wong-Baker FACES Pain Rating Scale, according to patient preference and age. For both scales, 0 corresponds with no pain and 10 corresponds with the highest pain.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Nasr, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bikmoradi A, Khaleghverdi M, Seddighi I, Moradkhani S, Soltanian A, Cheraghi F. Effect of inhalation aromatherapy with lavender essence on pain associated with intravenous catheter insertion in preschool children: A quasi-experimental study. Complement Ther Clin Pract. 2017 Aug;28:85-91. doi: 10.1016/j.ctcp.2017.05.008. Epub 2017 May 24. PMID 28779942
- [Result] Ghaderi F, Solhjou N. The effects of lavender aromatherapy on stress and pain perception in children during dental treatment: A randomized clinical trial. Complement Ther Clin Pract. 2020 Aug;40:101182. doi: 10.1016/j.ctcp.2020.101182. Epub 2020 Apr 28. PMID 32891272
- [Result] Kang HJ, Nam ES, Lee Y, Kim M. How Strong is the Evidence for the Anxiolytic Efficacy of Lavender?: Systematic Review and Meta-analysis of Randomized Controlled Trials. Asian Nurs Res (Korean Soc Nurs Sci). 2019 Dec;13(5):295-305. doi: 10.1016/j.anr.2019.11.003. Epub 2019 Nov 16. PMID 31743795
- [Result] Karaman T, Karaman S, Dogru S, Tapar H, Sahin A, Suren M, Arici S, Kaya Z. Evaluating the efficacy of lavender aromatherapy on peripheral venous cannulation pain and anxiety: A prospective, randomized study. Complement Ther Clin Pract. 2016 May;23:64-8. doi: 10.1016/j.ctcp.2016.03.008. Epub 2016 Mar 25. PMID 27157961
- [Result] Kucuk Alemdar D, Yaman Aktas Y. The Use of the Buzzy, Jet Lidokaine, Bubble-blowing and Aromatherapy for Reducing Pediatric Pain, Stress and Fear Associated with Phlebotomy. J Pediatr Nurs. 2019 Mar-Apr;45:e64-e72. doi: 10.1016/j.pedn.2019.01.010. Epub 2019 Jan 30. PMID 30711327